## **Mindfully Attending to Pain Sensations**

May 2, 2019

#### Informed Consent

Study Title: Mindfully Attending to Pain Experiences

Researchers: Katherine Bercovitz, Noga Tsur, Karyn Gunnet-Shoval, Ellen Langer

## **Participation is voluntary**

It is your choice whether or not to participate in this research. If you choose to participate, you may change your mind and leave the study at any time. Refusal to participate or stopping your participation will involve no penalty or loss of benefits to which you are otherwise entitled.

## What is the purpose of this research?

The purpose of this research is to assess the effects of monitoring pain symptoms through the use of mindfulness techniques in individuals experiencing chronic pain.

## How long will I take part in this research?

The bulk of your study participation will occur over a one-week period, with the opportunity to complete two brief follow-up surveys 1 month and 3 months later.

## What can I expect if I take part in this research?

### Online Questionnaires:

If you decide to participate, we will ask you to complete four online questionnaires (1 hour for the first and 30 minutes for each of the next three; Total time = 2.5 hours). These questions will ask you about demographics, pain history and experiences, mood, personality, mental health, day-to-day functioning, and feedback about the mindfulness exercises you will complete. We may text you to remind you of these surveys. If you receive these reminder text messages and no longer wish to receive them, you can let us know via text or email and we will stop sending them.

#### Daily Activities:

Every participant will be randomly assigned to one of three groups. This means that you have an equal chance of being in each group.

All participants will be asked to complete short at-home activities for one week. Participants will either be asked to complete one or multiple of the following activity components: a) daily mindfulness instructions; b) prompts to notice and report on your pain experience, c) prompts to notice your current activity. Your total at-home participation for the study will take anywhere from 30-60 minutes in total (5-15 minutes per day for 6 days).

## What are the risks and possible discomforts?

If you choose to participate, we do not anticipate risk beyond that which is minimal. Minimal psychological discomfort may occur, for example, as a result of reflecting on your pain experience or stress levels. Additionally, there is a chance that paying attention to pain sensations may cause people to feel more pain as a result of this increased attention. There is also a risk of answering text messages while operating heavy machinery or otherwise engaged. Finally, there is the risk that individuals may incur financial cost from receiving text

messages if they do not have an unlimited text messaging plan; we ask you to consider not participating in the study if you are concerned about having to pay extra text messaging costs.

To minimize these risks, you will be given a list of psychosocial resources at the start of the study for you to reference in the event that such discomfort(s) occur. Further, we provide our contact information in this Informed Consent should any concerns, at all, arise. We will also remind you not to answer our text messages prompts while operating heavy machinery or otherwise engaged.

## Possible benefits of being in this research study:

We cannot promise any benefits to you or others from your taking part in this research. However, possible benefits include improved wellbeing and increased knowledge about yourself. As stated above, our goal is to identify useful exercises for a future intervention that may help others suffering from chronic pain, so there are potential benefits for them as well.

## Will I be compensated for participating in this research?

You will will be entered into a raffle for a \$100 Amazon gift card upon completion of each online survey, with the opportunity to win up to \$400 in total gift card compensation. You have a 1/180 chance of winning one of these gift cards. In addition, you will receive a \$10 electronic gift card to either Amazon.com for completing the final survey.

# If I take part in this research, how will my privacy be protected? What happens to the information you collect?

The responses in the surveys will not be identified by your name or email address. If you would like to enter the raffle or receive a copy of the results of this study, you have the option to submit your email address, which will be retained on a password-protected computer until the results of the study are sent to you. Unless you specify that you would like us to retain this contact information in case of future study opportunities, it will be permanently deleted from the computer. All data will be published in aggregate.

# If I have any questions, concerns or complaints about this research study, whom can I talk to?

The researchers for this study are Katherine Bercovitz, Noga Tsur and Karyn Gunnet-Shoval who can be reached at kbercovitz@g.harvard.edu. The faculty sponsor is Ellen Langer who can be reached at 617-495-3860, and langer@wjh.harvard.edu.

- If you have questions, concerns, or complaints,
- If you would like to talk to the research team,
- If you think the research has harmed you, or
- If you wish to withdraw from the study.

This research has been reviewed by the Committee on the Use of Human Subjects in Research at Harvard University. They can be reached at 617-496-2847, Smith Campus Center, 1350 Massachusetts Avenue, Suite 935, Cambridge, MA 02138, or cuhs@harvard.edu for any of the following:

- If your questions, concerns, or complaints are not being answered by the research team,
- If you cannot reach the research team,
- If you want to talk to someone besides the research team, or
- If you have questions about your rights as a research participant.

## **Statement of Consent**

I have read the information in this consent form. All my questions about the research have been answered to my satisfaction.

## SIGNATURE

| Your signature below indicates your permission to take part in this provided with a copy of this consent form. | research. You will be |
|---|---|
| Printed name of participant | |
| Signature of participant | Date |